CLINICAL TRIAL: NCT04991649
Title: Effects of Acceptance and Commitment Therapy-based Asthma Management Training Program for Parents of Young Children With Neurodevelopmental Comorbidities: A Randomized Controlled Trial
Brief Title: ACT for Parents of Children With Neurodevelopmental Comorbidities
Acronym: ACTparenting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Yuen Yu CHONG, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07181086
Record Dates: First submitted 2021-08-01; First posted 2021-08-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Asthma in Children; Attention Deficit Hyperactivity Disorder
Keywords: Acceptance and Commitment Therapy; Asthma; Attention Deficit Hyperactivity Disorder; Randomized Controlled Trial
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Asthma

STUDY DESIGN:
Intervention Model Description: Parallel Assignment; repeated-measures 2-arm randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors and researchers (and health care staff of the study hospital) are blind to the group assignment and intervention undertaken and concealed to the participant list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT Group (Experimental): One two-weekly 2-hour of positive parenting program plus a four-weekly 2-hour group ACT program and routine pediatric asthma out-patient services, including medical follow-up, asthma education by Advanced Practice Nurse specialized in pediatric respiratory care, and referrals to community care/welfare by psychiatrist/medical social worker for parental training in ADHD care.
  Interventions: Behavioral: Acceptance and Commitment Therapy-based Asthma Management Training Program
- Treatment-as-usual (TAU) Group (Other): Routine pediatric asthma out-patient services, including medical follow-up, asthma education by Advanced Practice Nurse specialized in pediatric respiratory care, and referrals to community care/welfare by psychiatrist/medical social worker for parental training in ADHD care.
  Interventions: Behavioral: Treatment-as-usual Group

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy-based Asthma Management Training Program — In addition to the routine pediatric asthma outpatient service as received with the TAU group, participants in the ACT group will additionally receive a two-weekly 2-hour Positive Parenting Program (Triple-P) and a four-weekly 2-hour ACT program (a total of six weekly sessions, 6-8 parents per group). The Triple-P aims to increase parental self-regulation and positive parenting practices to promote child cooperation, lead to consistent discipline and promote routines in childhood asthma management. On the other hand, The ACT sessions foster parents' psychological flexibility to cultivate non-judgmental acceptance of difficult parenting experiences, be mindful in daily parenting, develop an observer-self, and promote commitment to one's values.
  Other Names: ACT Group
  Arms: ACT Group
Behavioral: Treatment-as-usual Group — Participants in the treatment-as-usual (TAU) group will receive routine pediatric asthma outpatient services. These services include regular follow-up appointments once every 3-6 months for reviewing the child's health conditions by pediatricians, refilling medications and asthma education (1.5-2 hours every 3-4 weeks) by Advanced Practice Nurse specialized in pediatric respiratory care, and referrals to community care/welfare services by psychiatrist/medical social worker for parental training in ADHD care.
  Other Names: TAU Group
  Arms: Treatment-as-usual (TAU) Group

SUMMARY:
This randomized controlled trial aims to examine the effectiveness of the Acceptance and Commitment Therapy-based Asthma Management Training Program on the health outcomes of asthmatic children with attention deficit hyperactivity disorder (ADHD) and their caregivers over a 12-month post-intervention.

DETAILED DESCRIPTION:
Background: Attention deficit hyperactivity disorder and asthma are two of the most common pediatric chronic conditions. A meta-analysis of 49 datasets worldwide and a population-based cohort analysis of 1.5 million individuals showed an adjusted OR of 1.6 for ADHD during school years if the child has asthma at early childhood. Multiple mechanisms underlying this temporal association have been suggested, including the impacts of inflammatory mechanism or immune dysregulation on brain development, as well as the chronic sleep disruption after allergic symptoms. Compared with children with only asthma, asthmatic children with neurodevelopmental diseases have a higher risk of emergency care visits due to an asthma attack (adjusted prevalence = 1.5). Although the exact mechanism is still unclear, it has been shown that parents' psychological difficulties play an influential role in the cascade of family, biological and psychological influences on children's asthma. Compared with non-ADHD families, parents of children with ADHD have higher parenting stress, and the risk of depression/anxiety is almost tripled. Due to parental distress, these parents may weaken their motivation and coping ability to manage childhood asthma, leading to poor asthma outcomes.

Although studies have shown that asthma education and parental programs are effective ways to improve asthma management skills and parenting skills, none of these interventions addresses the psychological needs of parents when dealing with children with ADHD. This study is a randomized controlled trial designed to examine the effectiveness of the family-based asthma management program in Hong Kong that uses Acceptance and Commitment Therapy (ACT) in fostering parents' psychological flexibility, bettering their psychological difficulties acceptance, and striving toward values-based goals to healthy functioning. It is expected that the ACT-based asthma management training program can help parents to be aware of their emotional state when interacting with asthmatic children with ADHD enabling them to effectively implement the children's asthma management and parenting skills they have learned, leading to the ultimate improvement of children's health outcomes. If it is found that the plan can effectively improve their lives by addressing the unmet psychological needs of parents of asthmatic children with ADHD, it can be incorporated into existing services in hospitals and community settings in Hong Kong and other Chinese communities.

Aim and hypothesis to be tested: When compared with the treatment-as-usual group, participants in the ACT-based Asthma Management Training Program will:

1. reduce asthmatic children' unscheduled visits due to his/her asthma exacerbations,
2. reduce asthmatic children' asthma symptoms,
3. reduce asthmatic children' ADHD symptoms,
4. reduce asthmatic children' asthma-related behavioral problems,
5. improve asthmatic children' caregivers' psychological flexibility and adjustment,
6. enhance parenting competence, parental asthma management self-efficacy, and parental and family functioning

Design: An randomized controlled trial with a two-arm and repeated-measures design

Participants: 118 Cantonese-speaking asthmatic children aged 3 - 12 years old with ADHD condition and their primary caregiver.

Instruments: Validated questionnaires

Interventions: The ACT-based Asthma Management Training Program consists of a two-weekly group Positive Parenting Program (Triple-P) workshop and a four-weekly group Acceptance and Commitment Therapy (ACT) program.

Primary outcome measure: Children's unplanned health care service visits due to asthma exacerbations over 12 months

Expected results: After participating in the ACT-based asthma management program, parents will become more psychologically flexible in caring for children with asthma comorbid with ADHD. Parents also acquire better parenting competence and children's asthma management skills, improving parental and family functioning and child health outcomes.:

ELIGIBILITY:
Inclusion Criteria:

* Children between the age 3 and 12
* Age of the child's primary caregiver between the age 18 and 65
* Diagnosed as asthma by a physician (ICD-10 codes J45, J46) as documented in his/her medical records as well as reported score more or equal 19 in the Childhood Asthma Control Test (C-CAT, or Asthma Control Test for child aged 12) indicating not well-controlled.
* Co-occur with a diagnosis with the attention deficit and hyperactivity disorder (ADHD) as documented in the patient history profile of the medical record by a child psychiatrist/medical doctor according to the criteria set forth by the Diagnostic and Statistical Manual of Mental Disorders (5th ed.; American Psychiatric Association [APA], 2013) or ICD-10.

Exclusion Criteria:

* Participant and/or his/her primary caregiver currently participate in another asthma-related intervention study
* Participant is under the care due to significant medical morbidities, including congenital problems, oxygen-dependent conditions, or the presence of a tracheotomy

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2021-04-11 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
The frequency of the unscheduled childhood asthma exacerbations visits | Change from baseline assessment to 12 months post-intervention
  The frequency of unscheduled healthcare service visits due to asthma exacerbations, including the public/private hospital emergency department visits, general outpatient clinic visits and private practitioners' clinic visits, hospital admission, and hospital stay length, will be collected by retrieving their medical records. A lessened frequency of unscheduled childhood asthma exacerbations visits signifies improved prevention and management of asthma cases. Any data (especially related to private healthcare services) that cannot be retrieved by the aforementioned method will be collected through parent-report questionnaires over 12 months.

SECONDARY OUTCOMES:
Child's asthma symptoms | Change from baseline assessment to 12 months post-intervention
  The 7-item Chinese Version of Childhood Asthma Control Test (C-CACT; Chen et al., 2008) is based on the Global Asthma Initiative clinical guidelines to assess the level of asthma control in children clinically. The C-CACT is divided into two parts. The first part is rated by the child on his/her own or with the caregiver's guidance consisting of 4 response options on the perception of asthma control, limitation of activities, coughing, and awakenings at night. Each question of the first part has four options from 0 to 3. The second part of the questionnaire is filled by the parent or the primary caregiver consisting of 3 questions, including reporting daytime symptoms, daytime wheezing, and night awakenings, using a 6-point Likert scale from 0 (Everyday) to 5 (Not at all). The sum of all scores yields the total score ranging from 0 to 27, with higher scores indicating greater asthma control. A score less than 20 shows inadequately controlled asthma.
Child's asthma-related behavioral problems | Change from baseline assessment to 12 months post-intervention
  The Asthma Behavior Checklist (ABC; Morawska, Stelzer, & Burgess, 2008) consists of 22 behaviors that parents with asthmatic children often have to manage and will be used to assess the degree of behavioral problems associated with asthma. Parents will provide each item with a score for his/her child's asthma-related behavioral problem, using a 7-point Likert scale, ranging from 1 (Not at all) to 7 (Very much) (ABC degree α=.93). Add all the 22 items together to get the total score. The higher the score, the more child's behavioral difficulties associated with asthma.
Child's ADHD symptoms | Change from baseline assessment to 12 months post-intervention
  The 18-item Chinese Strengths and Weaknesses of ADHD-symptoms and Normal-Behavior (Chinese SWAN; Lai et al., 2013) will be used to measure the child's ability to focus attention, control activity, and inhibit impulses. SWAN is developed based on the DSM-IV standard of ADHD and has high sensitivity and specificity (clinical cut-off value >90%). Parents rated the items on a 7-point response scale (-3 = far above average; -2 = above average; -1 = somewhat above average; 0 = average; 1 = somewhat below average; 2 = below average; 3 = far below average). The mean score of all the 18 items provides the ADHD-Combined (ADHD-C) score, whereas Questions 1 to 9 constitute the ADHD-Inattentive (ADHD-I) score, and Questions 10 to 18 the ADHD-Hyperactivity/Impulsivity (ADHD-HI) score. According to their respective scales or subscales, higher scores indicate higher levels of ADHD symptoms or problem behaviors.
Parent's psychological flexibility | Change from baseline assessment to 12 months post-intervention
  The 7-item Chinese version of the Acceptance and Action Questionnaire-II (AAQ-II; Chong et al., 2019) will be used to measure the participating parents' psychological inflexibility, the dominance of internal events over contingencies in determining value-directed actions preventing people from making full contact with the present moments. A 7-point Likert scale is used, ranging from 1 (never true) to 7 (always true). The item scores are added together to create a total score (range 7 to 49). The higher the total score, the poor psychological flexibility (more psychologically inflexible), and the lower the total score, the better the psychological flexibility. The AAQ-II demonstrated good internal consistencies (α = .88) and test-retest reliabilities (r = .79 - .81) among the Hong Kong adult population.
Parent's psychological adjustment to the child's illness | Change from baseline assessment to 12 months post-intervention
  The 25-item Chinese Version of Parent Experience of Child Illness (PECI; Chong et al., 2019) scale will be used to capture the psychological adjustment of parents in caring for a child with chronic diseases on a 5-point Likert scale ranging from 0 (never) to 4 (always), with two scales, PECI Distress Scale (consisting of 3 subscales: Guilt and Worry, Unresolved Sorrow and Anger, and Long-term Uncertainty) and PECI Resources Scale (consisting of 1 subscale: Emotional Resources). The scores of each subscale are added and then divided by the number of items. The PECI Distress Score and Resources Score evaluate the distress and perceived resources of caregivers of children suffering from chronic diseases. Each PECI score had adequate internal consistencies (α=.72-.89) and test-retest reliabilities (r=.83-.86) in HK parents of children with asthma.
Parent's parenting competence | Change from baseline assessment to 12 months post-intervention
  The 17-item Chinese Version of the Parenting Sense of Competency Scale (C-PSOC; Ngai, Chan,& Holroyd E, 2007) will be used to assess parents' perceptions of their abilities to manage parenting needs. The PSOC comprises two subscales - the Efficacy subscale, and the Satisfaction subscale. The Efficacy subscale contains eight items measuring parents' perception of competence in the parenting role. Differently, the Satisfaction subscale contains nine items evaluating the satisfaction and comfort of parents with the parenting role. Each item is scored using a 6-point Likert scale, ranging from 1 (strongly disagree) to 6 (strongly agree). The total score ranges from 17 to 102, while subscale scores range for the Efficacy and Satisfaction subscales are 17 to 48 and 17 to 54, respectively. The higher the score, the higher sense of competence and satisfaction in parenting. The PSOC had adequate internal consistencies (α=.77-.85) and test-retest reliabilities (r=.87) among Hong Kong parents.
Parent's asthma management self-efficacy | Change from baseline assessment to 12 months post-intervention
  The 13-item Chinese Version of Parent Asthma Management Self-Efficacy (PAMSE; Chong et al., 2019) scale will be employed to assess parents' self-efficacy in preventing and managing childhood acute asthma exacerbations, using a 5-point Likert scale from 1 (not at all sure) to 5 (completely sure). The PAMSE comprises two subscales that measure attack prevention self-efficacy (6 items) and attack management self-efficacy (7 items). All scores are calculated by adding up all items and dividing by the number of items. A higher score indicates better self-efficacy in the respective scales. The PAMSE had adequate internal consistencies (α=.77 - .82) and test-retest reliabilities (ICC=.76 - .87) in Hong Kong parents of children with asthma.
Parental and family functioning | Change from baseline assessment to 12 months post-intervention
  The 36-item Chinese version of the Pediatric Quality of Life Inventory Family Impact Module (PedsQL FIM; Chen et al., 2011) will be adopted to assess the impact of pediatric asthma comorbid with ADHD on parent health-related quality of life and the family functioning. The PedsQL FIM consists of 8 subscales: Physical Functioning (6 items), Emotional Functioning (5 items), Social Functioning (4 items), Cognitive Functioning (5 items), Communication (3 items), Worry (5 items), Daily Activities (3 items) and Family Relationships (5 items). The former six subscales measure parents' overall functioning, while the latter two subscales measure parent-reported family functioning. Each item has five Likert response options, which are 0 (never a problem) to 4 (almost always a problem). Items are then linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0) and averaged by the number of items, so that higher scores indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yuen Yu CHONG, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Paediatrics and Adolescent Medicine, Tuen Mun Hospital, Tuenmen, Hong Kong

REFERENCES:
- [Derived] Chong YY, Chien WT, Fung KP, Leung SP, Lam SY. Acceptance and Commitment Therapy-Based Parenting Program in Children With Co-Occurring Asthma and ADHD: A Randomized Clinical Trial. JAMA Pediatr. 2025 Aug 1;179(8):846-856. doi: 10.1001/jamapediatrics.2025.1313. PMID 40455452